CLINICAL TRIAL: NCT06695247
Title: Mobility Outcomes in Post-Pulmonary Embolic Disease (MOPED): A Pilot Feasibility Prospective Randomized Trial
Brief Title: A Study of Mobility Outcomes in Post-Pulmonary Embolic Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stan Henkin, Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-009493
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-Based Exercise Training (Experimental)
  Interventions: Other: Exercise Training
- Standard therapy (Standard of Care) (No Intervention)

INTERVENTIONS:
Other: Exercise Training — Patients will be recommended to exercise 3 days/week, 20 minutes per session, for 12 weeks using personalized intervention determined by a consultation with a clinical exercise physiologist (CEP)
  Arms: Home-Based Exercise Training

SUMMARY:
The purpose of this study is to develop a unique structure and delivery of home-based exercise through multidisciplinary expertise of cardiovascular medicine specialists and cardiac physiologists using an Interactive Care Plan.

ELIGIBILITY:
Inclusion Criteria:

Acute intermediate-risk PE, defined as:

* Intraluminal filling defect in segmental or larger vessels on computed tomography pulmonary angiography or high-probability ventilation/perfusion scan AND
* Evidence of right ventricular enlargement by computed tomography (RV to LV ratio >1) or echocardiography; and/or right ventricular dysfunction by transthoracic echocardiography. These imaging characteristics must be in the setting of acute PE rather than explained by a prior chronic condition.

Acute high-risk PE, defined as:

* Intraluminal filling defect in segmental or larger vessels on computed tomography pulmonary angiography or high-probability ventilation/perfusion scan AND
* Evidence of right ventricular enlargement by computed tomography (RV to LV ratio >1) or echocardiography; and/or right ventricular dysfunction by transthoracic echocardiography. These imaging characteristics must be in the setting of acute PE rather than explained by a prior chronic condition; AND
* Hypotension (systolic blood pressure < 90 mm Hg sustained for more than 15 minutes; or requiring vasopressors) or cardiogenic shock due to acute pulmonary embolism.

Exclusion Criteria:

* Inability to ambulate independently, which is necessary to perform 6MWD (may be self-reported or as deemed by physical therapy during inpatient evaluation).
* If patient requires supplemental oxygen during ambulation, this does not exclude patient from participation and will be noted during eCRF.
* Prior history of pulmonary embolism
* History of CTEPH or pulmonary arterial hypertension
* Unable to read a questionnaire in English
* Unable to return for baseline, 3- or 6-month follow-up visit
* Pregnancy-associated pulmonary embolism
* Life expectancy <1 year based on comorbidities
* Unable/unwilling to provide informed written consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in physical capacity from baseline | Baseline, 3 Months, 6 Months
  Physical capacity will be determined by 6-minute walk distance (6MWD)

SECONDARY OUTCOMES:
Change in Pulmonary Embolism-specific quality of life (PEmb-QOL) outcome measures from baseline | Baseline, 3 Months, 6 Months
  The Pulmonary Embolism-specific quality of life questionnaire assesses 6 quality of life dimensions in individuals with history of PE: frequency of symptoms, intensity of symptoms, activities of daily living limitations, social limitations, emotional distress, and work-related problems. Higher scores indicate worse quality of life.
Change in general Short Form 36 (SF-36) quality of life outcome measures from baseline | Baseline, 3 Months, 6 Months
  The Short Form 36 (SF-36) questionnaire assesses 8 quality of life dimensions: physical activity limitations, social activities limitations, activities of daily living physical limitations, bodily pain, general mental health, activities of daily living emotional limitations, vitality, and general health perceptions. Higher scores indicate better quality of life.
Number of Steps | Baseline, 3 Months, 6 Months
  Number of Steps will be determined by fitbit tracking with Fitabase.

CONTACTS AND LOCATIONS:
Overall Officials: Stan Henkin, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No